CLINICAL TRIAL: NCT01517919
Title: Peer-Led Self-Management Support in "Real World" Clinical and Community Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: American Academy of Family Physicians (Other)
Responsible Party: Principal Investigator, Rebecca Mase, Michele Heisler, MD, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DRDA 90-0893
Record Dates: First submitted 2012-01-17; First posted 2012-01-25 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Diabetes
Keywords: peer support; peer leader; community health worker; empowerment; self-management
MeSH Terms: conditions — Diabetes Mellitus; Empowerment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention: Peer Led Self-Management (Experimental): Intervention: Peer Led Self-Management (PLSM) involves the DSME program followed by 12 months of peer-led ongoing self-management support
  Interventions: Behavioral: Peer-Led Self-Management
- Diabetes Self-Management Education (No Intervention): Control: Diabetes Self-Management Education (DSME) involves 12 sessions of self-management training including diabetes education, one-on-one sessions, bi-weekly phone contacts, and preparation for a clinic visit.

INTERVENTIONS:
Behavioral: Peer-Led Self-Management — The PLSM intervention is designed to improve and sustain participants' self-management and health-related gains associated with type 2 diabetes. The role of peer leaders is to provide support for (1) ongoing self-management efforts (including the 5-step "action-planning" process), (2) psychosocial and emotional adjustment, and (3) linkage to needed health care resources.
  PLSM intervention will consist of three main components provided by the Peer Leaders: weekly self-management support sessions; outreach telephone contacts and inbound telephone call from participants.
  Other Names: Peer Leadership; Peer Support
  Arms: Intervention: Peer Led Self-Management

SUMMARY:
This study will systematically evaluate a training program in state-of-the-art behavioral change approaches and facilitation skills for peer leaders and a peer-led diabetes self-management support program designed to be conducted in community and clinic-based settings on an ongoing basis.

DETAILED DESCRIPTION:
In phase one we will develop and evaluate a theoretically-driven program to train peer leaders to facilitate longer-term empowerment-based interventions that, when led by health care professionals, have been associated with improved diabetes-related health and psychosocial outcomes.1-8 In phase two we will examine the impact of a sustained peer-led, empowerment-based self-management intervention on improving and maintaining diabetes-related health outcomes. We propose to develop and test the training and program simultaneously in two distinct cultural and linguistic communities with which the team already has strong working relationships and a track record of prior work: African-American (AA) adults in a community-based setting (Ypsilanti, Michigan) and Latino adults (Spanish- and English-speaking) in a clinic-based setting (Southwest Detroit). This will allow us to compare and contrast the translations of the training and program in these two different contexts and to better refine and understand effective methods and develop culturally tailored training and program materials in both English and Spanish.

ELIGIBILITY:
Inclusion Criteria:

* the study will recruit African Americans and Latinos with type 2 diabetes, - at least 21 years old, and
* who have a regular health care provider, and
* will commit to attend the 12 session DSME program.

Exclusion Criteria:

* having physical limitations preventing participation, and
* other serious health conditions (e.g., terminal cancer),
* serious psychiatric illness, self-reported excessive alcohol or illicit drug use, and
* serious diabetes complications (e.g., blindness) that would impede meaningful participation in the program

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2010-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Changes in clinical, self-care and diabetes-related quality of life from baseline | Measured at completion of 12 session DSME program, DSME program completion occurs between 3 and 6 months following enrollment; 6 months post-completion; 12 months post-completion
  Clinical, self-care and diabetes-related quality of life improvements including the following measures: A1c, Summary of Diabetes Self-Care Activities Measure, Diabetes Distress Scale (DDS)

SECONDARY OUTCOMES:
Changes in clinical, self-care and diabetes-related quality of life from baseline | Measured at completion of 12 session DSME program, DSME program completion occurs between 3 and 6 months following enrollment; 6 months post-completion; 12 months post completion
  Clinical, self-care and diabetes-related quality of life improvements including the following measures: lipid levels, blood pressure reading, height and weight, BMI, and satisfaction with care.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Heisler, MD, MPA, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States